CLINICAL TRIAL: NCT06168253
Title: Text Message Safety Behavior Fading Intervention for Social Anxiety
Brief Title: Text Message Safety Behavior Fading for Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY2247MOD4140
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Social Anxiety
Keywords: Social Anxiety; Safety Behaviors; Intervention; Text-message

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in to one of two conditions
Who Masked: Participant
Masking Description: Participants will receive one of two matched interventions. They will not be told whether they are receiving the active or control intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Safety Behavior Fading (Experimental): This treatment lasts a total of 28 days. Participants will be asked to identify common safety behaviors related to social anxiety. For the next 14 days, participants will receive instructions to fade out these behaviors. After 14 days, participants will be asked to re-select their target safety behaviors and continue to reduce them over the next two weeks.
  Interventions: Behavioral: Safety Behavior Fading for Social Anxiety
- Unhealthy Behavior Fading (Active Comparator): This treatment lasts a total of 28 days. Participants will be asked to identify common unhealthy behaviors related to social anxiety. For the next 14 days, participants will receive instructions to fade out these behaviors. After 14 days, participants will be asked to re-select their target unhealthy behaviors and continue to reduce them over the next two weeks.
  Interventions: Behavioral: Unhealthy Behavior Fading

INTERVENTIONS:
Behavioral: Safety Behavior Fading for Social Anxiety — Participants are asked to reduce or eliminate safety behaviors via text message reminders and checklists to monitor progress.
  Arms: Experimental: Safety Behavior Fading
Behavioral: Unhealthy Behavior Fading — Participants are asked to reduce or eliminate unhealthy behaviors via text message reminders and checklists to monitor progress.
  Arms: Unhealthy Behavior Fading

SUMMARY:
The current study aims to explore the efficacy of a text message based Safety Behavior Fading Intervention compared to an active control intervention.

DETAILED DESCRIPTION:
Safety behavior fading may be a viable standalone intervention for social anxiety. In the present trial, participants high in social anxiety will be randomized to either receive a daily checklist exercise aimed at eliminating (1) safety behaviors or (2) unhealthy behaviors. Individuals randomly assigned to the safety behavior fading condition will receive instructions to decrease or eliminate their four most habitual social anxiety safety behaviors. In addition, they will receive daily reminders via text message to decrease these behaviors, along with a safety behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each safety behavior over the previous day. Individuals randomly assigned to the control condition will receive similar text messages and a daily checklist to encourage fading of unhealthy behaviors. Participants in both conditions will complete checklists for 28 days. After day 14 of treatment, participants will re-select their target safety behaviors or unhealthy behaviors, and will then be prompted to reduce these new behaviors for another 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Social Phobia Inventory Score >29
* Stable Psychotropic Medications for 4 weeks prior to participation

Exclusion Criteria:

* Currently participating in psychotherapy for social anxiety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Social Phobia Inventory (SPIN) | Time Frame: Day 0, Day 14, Day 28, Day 56
  Self-report scale that measures Social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety symptoms.

SECONDARY OUTCOMES:
Change in Center For Epidemiological Studies Depression Scale, Ten Item Version (CESD-10) | Time Frame: Day 0, Day 28, Day 56
  A 10-item self-report scale measuring depression symptoms; higher scores indicate greater depressive symptoms.
Change in UCLA Loneliness Scale, Short Form (ULS-8) | Time Frame: Day 0, Day 28, Day 56
  An 8-item self-report measure of subjective loneliness, with higher scores indicating greater loneliness.
Change in Self-Beliefs Related to Social Anxiety Scale (SBSA) | Time Frame: Day 0, Day 28, Day 56
  A 15-item scale measuring common and generally maladaptive beliefs related to social anxiety.
Change in Subtle Avoidance Frequency Examination (SAFE) scale | Time Frame: Day 0, Day 28, Day 56
  A 32-item self-report measure of safety behavior usage frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No